CLINICAL TRIAL: NCT06829745
Title: The Effect of Laughter Yoga Practiced After Burn Dressing on Pain, Anxiety and Mental Well-Being Levels.
Brief Title: The Effect of Laughter Yoga Practiced After Burn Dressing
Acronym: laughteryoga
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Fatma Özdemir Şahin, principal Investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SBÜ-HEM-FOŞ-01
Record Dates: First submitted 2025-02-06; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Burns; Laughter Yoga
Keywords: Burns; Laughter Yoga
MeSH Terms: conditions — Burns | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: It is a prospective interventional type two-group randomized controlled clinical study. Distribution according to the groups and layers to be assigned for each intervention; Group-1 (Experiment) was designed as clinical routine (Laughter yoga), and Group-2 (Control) was designed as clinical routine.
Masking Description: When laughter yoga studies in the literature are examined, the laughter yoga practitioner is the researcher himself. Therefore, due to the nature of the application method to be used, the patients and the researcher are not considered blind. The evaluator will be considered blind in the analysis of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1(Laughter Yoga) (Experimental): Group-1(Laughter Yoga) Data will be obtained through the Introductory Information Form, Visual Analogue Scale (VAS), State Anxiety Scale and Warwick Edinburgh Mental Well-Being Scale. Patients who will receive burn dressing will be visited in the clinic before the dressing and will be informed about the study. Sampled individuals will be placed into intervention and control groups using a random number table created with MS Excel software. The average hospital stay of patients is three weeks. Within the scope of the study, laughter yoga will be applied 2 hours after the dressing to the patients who are treated in the burn clinic for three weeks and are included in the intervention group(30 minutes).
  Interventions: Other: Laughter Yoga
- Group 2 (Clinical routine) (No Intervention): For the control group, STAII State Anxiety Scale, Visual Analog Scale (VAS) and Warwick Edinburgh Mental Well-Being Scale levels will be determined in the same periods without any application.

INTERVENTIONS:
Other: Laughter Yoga — Laughter yoga is applied to the intervention group patient 2 hours after the burn dressing. It is applied every other day for 30 minutes after dressing for three weeks.
  Arms: Group 1(Laughter Yoga)

SUMMARY:
Burn is a serious trauma that causes acute damage to the skin and subcutaneous tissues due to the effect of heat, electricity, radiation, physical, and chemical substances. Research shows a relationship between burn dressing changes and increased pain, anxiety, and stress. It can also be said that anxiety negatively affects wound healing. This study aimed to determine the effect of Laughter Yoga, a non-drug method, on reducing or completely eliminating pain and anxiety after burn dressing and increasing the level of mental well-being. This study is planned to be conducted in a randomized manner.

DETAILED DESCRIPTION:
The Burn Center will consist of patients receiving treatment at the Burn Clinic. Data will be obtained through the Introductory Information Form, Visual Analogue Scale (VAS), State Anxiety Scale and Warwick Edinburgh Mental Well-Being Scale. Patients who will receive burn dressing will be visited in the clinic before the dressing and will be informed about the study. Sampled individuals will be placed into intervention and control groups using a random number table created with MS Excel software. The average hospital stay of patients is three weeks. Within the scope of the study, laughter yoga will be applied 2 hours after the dressing to the patients who are treated in the burn clinic for three weeks and are included in the intervention group.

For the control group, STAII State Anxiety Scale, Visual Analog Scale (VAS) and Warwick Edinburgh Mental Well-Being Scale levels will be determined in the same periods without any application. The data obtained will be analyzed with appropriate statistical methods using the SPSS for Windows 23.0 program (Statistical Package for the Social Sciences).

ELIGIBILITY:
Inclusion Criteria:

* Receiving inpatient treatment in hospital due to burns,
* Between the ages of 18 and 60, (sick individuals over the age of 60 may have chronic diseases and have problems complying with commands)
* Those with moderate or large severity burns (according to the Turkish Ministry of Health, Burn Injury Treatment Algorithm (11)).
* In individuals with 2nd degree burns, the total burn width does not exceed 40%, and in those with 3rd degree burns, the total burn width does not exceed 10%,
* At least 2 days have passed since the burn injury (the inflammatory phase has passed during the wound healing process and is in the proliferation phase),
* Not in the maturation phase according to the wound healing process, No burns in the abdomen and head and neck area (due to preventing the possible negative effects of Laughter Yoga on the specified areas)
* Patients who volunteer to participate in the research will be included in the study.

Exclusion Criteria:

* Using anxiolytic and sedative drugs,
* Having a psychiatric illness,
* Patients with communication disabilities will not be included in the research.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Level of mental well-being | The mental well-being scale will be used 3 times in total: before dressing, after 3 weeks of laughter yoga, and 10 days after discharge.
  The emergence of mental well-being in the dimension consisting of 14 positive items. Scoring of the performance is on a 5-point Likert type, where 1 = I do not agree at all, 2 = I disagree, 3 = I somewhat agree, 4 = I configure, 5 = completely structured, and a minimum of 14 and a maximum of 70 points can be obtained from the dimension.
Visual Analogue Scale (VAS) for Pain and Satisfaction Levels | VAS will be taken before the laughter yoga practice. It will be taken after the laughter yoga practice. It will be repeated a total of 18 times, on sunburn dressing days, for 3 weeks.
  The Visual Analog Scale is a one-dimensional scale commonly used to measure pain intensity. VAS is a measuring tool with a length of 0-10 cm (0-100 mm). This measuring tool can be used horizontally or vertically. The scale starts with "no pain" and ends with "unbearable pain". High scores from the scale indicate high pain intensity. The cut-off points for pain scores taken from the scale are recommended as 0-4 mm "no pain", 5-44 mm "mild pain", 45-74 mm "moderate pain" and 75-100 mm "severe pain" (89). In our study, the VAS scale will be used horizontally and in cm to measure patients' pain intensity and satisfaction levels.
State-Trait Anxiety Inventory level | State-Trait Anxiety Inventory level will be taken before the laughter yoga application. It will be taken after the laughter yoga application. It will be repeated 18 times in total, on sunburn dressing days for 3 weeks.
  "State Anxiety Inventory (STAI-I)" is a tool that allows measuring how an individual feels at a certain moment and situation, that is, the level of anxiety in that situation. Each item in this inventory consists of four options: 1 (Not at all), 2 (Somewhat), 3 (Quite a bit), and 4 (Completely), which determine the intensity of the emotions felt by individuals at that moment.

CONTACTS AND LOCATIONS:
Overall Officials: fatma sahin, Principal Investigator — Kartal Dr. Lütfi Kırdar Şehir Hastanesi
Locations (2):
- Turkey (Türkiye) (2):
  - Dr. Lütfi Kırdar Şehir Hastanesi, Istanbul, Kartal
  - Kartal Dr. Lütfi Kırdar Şehir Hastanesi, Istanbul, Kartal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Han S, Zhang L, Li Q, Wang X, Lian S. The Effects of Laughter Yoga on Perceived Stress, Positive Psychological Capital, and Exercise Capacity in Lung Cancer Chemotherapy Patients: A Pilot Randomized Trial. Integr Cancer Ther. 2023 Jan-Dec;22:15347354231218271. doi: 10.1177/15347354231218271. PMID 38102816
- [Background] Morishima T, Miyashiro I, Inoue N, Kitasaka M, Akazawa T, Higeno A, Idota A, Sato A, Ohira T, Sakon M, Matsuura N. Effects of laughter therapy on quality of life in patients with cancer: An open-label, randomized controlled trial. PLoS One. 2019 Jun 27;14(6):e0219065. doi: 10.1371/journal.pone.0219065. eCollection 2019. PMID 31247017
- [Background] Hayashi K, Kawachi I, Ohira T, Kondo K, Shirai K, Kondo N. Laughter and Subjective Health Among Community-Dwelling Older People in Japan: Cross-Sectional Analysis of the Japan Gerontological Evaluation Study Cohort Data. J Nerv Ment Dis. 2015 Dec;203(12):934-942. doi: 10.1097/NMD.0000000000000399. PMID 26649930